CLINICAL TRIAL: NCT04712097
Title: Phase III Randomized, Open-Label, Multicenter Study Evaluating Efficacy and Safety of Mosunetuzumab in Combination With Lenalidomide in Comparison to Rituximab in Combination With Lenalidomide With a Non-Randomized Single Arm US Extension of Mosunetuzumab in Combination With Lenalidomide in Patients With Follicular Lymphoma After at Least One Line of Systemic Therapy
Brief Title: A Study Evaluating the Efficacy and Safety of Mosunetuzumab in Combination With Lenalidomide in Comparison to Rituximab in Combination With Lenalidomide With a US Extension of Mosunetuzumab in Combination With Lenalidomide in Participants With Follicular Lymphoma
Acronym: Celestimo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO42909; 2020-005239-53 (EudraCT Number)
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Follicular Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- M + Len (Arm A) (Experimental): Participants will receive mosunetuzumab for 12 cycles, plus lenalidomide from cycles 2-12 (Cycle length = 21 days for Cycle 1; cycle length = 28 days for Cycles 2-12)
  Interventions: Drug: Mosunetuzumab; Drug: Lenalidomide; Drug: Tociluzumab
- R + Len (Arm B) (Experimental): Participants will receive weekly rituximab in Cycle 1, then on Day 1 of Cycles 3, 5, 7, 9, and 11. Participants will also receive lenalidomide in Cycles 1-12. (Cycle length = 28 days for Cycles 1-12)
  Interventions: Drug: Lenalidomide; Drug: Rituximab; Drug: Tociluzumab
- M + Len (US Extension Arm C) (Experimental): Participants will receive mosunetuzumab for 12 cycles, plus lenalidomide from cycles 2-12 (Cycle length = 21 days for Cycle 1; cycle length = 28 days for Cycles 2-12)
  Interventions: Drug: Mosunetuzumab; Drug: Lenalidomide; Drug: Tociluzumab

INTERVENTIONS:
Drug: Mosunetuzumab — Participants will receive intravenous (IV) mosunetuzumab in a step-up dosing schedule on Days 1, 8, and 15 of Cycle 1, and on Day 1 of Cycles 2-12
  Arms: M + Len (Arm A); M + Len (US Extension Arm C)
Drug: Lenalidomide — Participants will receive oral lenalidomide once daily on Days 1-21 of Cycles 2-12 (M + Len) or Cycles 1-12 (R + Len)
Drug: Rituximab — Participants will receive IV rituximab on Days 1, 8, 15, and 22 of Cycle 1, then on Day 1 of Cycles 3, 5, 7, 9, and 11
  Arms: R + Len (Arm B)
Drug: Tociluzumab — Tocilizumab will be administered as needed to manage cytokine release syndrome (CRS) events

SUMMARY:
This study will evaluate the efficacy and safety of mosunetuzumab in combination with lenalidomide (M + Len) compared to rituximab in combination with lenalidomide (R + Len) in participants with relapsed or refractory (R/R) follicular lymphoma (FL) who have received at least one line of prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Histologically documented CD20+ FL (Grades 1-3a)
* Requiring systemic therapy assessed by investigator based on tumor size and/or Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria
* Received at least one prior systemic lymphoma therapy, which included prior immunotherapy or chemoimmunotherapy
* Availability of a representative tumor specimen and the corresponding pathology report at the time of relapse/persistence for confirmation of the diagnosis of FL. Pretreatment sample of at least 1 core-needle, excisional or incisional tumor biopsy is required. Cytological or fine-needle aspiration samples are not acceptable. Fresh pretreatment biopsy is preferred. Patients who are unable to undergo biopsy procedures may be eligible for study enrollment if an archival tumor tissue sample (preferably from the most recent relapse/persistence) as paraffin blocks or at least 15 unstained slides, or in accordance with local regulatory requirements, can be sent to the Sponsor.
* Adequate hematologic function (unless due to underlying lymphoma, per the investigator)
* Agreement to comply with all local requirements of the lenalidomide risk minimization plan, which includes the global pregnancy prevention program.
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use 2 adequate methods of contraception, including at least 1 method with a failure rate of < 1% per year, for at least 28 days prior to Day 1 of Cycle 1, during the treatment period (including periods of treatment interruption), and for at least 28 days after the last dose of lenalidomide, 3 months after the final dose of tocilizumab (if applicable), mosunetuzumab, and 12 months after final dose of rituximab. Women must refrain from donating eggs during this same period.
* For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 28 days after last dose of lenalidomide, 3 months after the final dose of tocilizumab (if applicable), mosunetuzumab and 12 months after the final dose of rituximab. Men must refrain from donating sperm during this same period.

Exclusion Criteria:

* Grade 3b FL
* Any history of disease transformation and/or diffuse-large B cell lymphoma (DLBCL)
* Documented refractoriness to lenalidomide, defined as no response (partial response or complete response) or relapse within 6 months of therapy
* Active or history of CNS lymphoma or leptomeningeal infiltration
* Prior standard or investigational anti-cancer therapy as specified: Lenalidomide exposure within 12 months prior to Day 1 of Cycle 1; Chimeric antigen receptor T cell therapy within 30 days prior to Day 1 of Cycle 1; Radioimmunoconjugate within 12 weeks prior to Day 1 of Cycle 1; Monoclonal antibody or antibody-drug conjugate within 4 weeks prior to Cycle 1 Day 1; Treatment with any anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first dose of study treatment
* Clinically significant toxicity (other than alopecia) from prior treatment that has not resolved to Grade </= 1 (per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0) prior to Day 1 of Cycle 1
* Treatment with systemic immunosuppressive medications, including, but not limited to prednisone (> 20 mg), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1
* History of solid organ transplantation
* History of severe allergic or anaphylactic reaction to humanized, chimeric or murine monoclonal antibodies
* Known sensitivity or allergy to murine products
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary (CHO) cells or any component of the mosunetuzumab, rituximab, tocilizumab, lenalidomide, or thalidomide formulation, including mannitol
* History of erythema multiforme, Grade >/= 3 rash, or blistering following prior treatment with immunomodulatory derivatives
* History of interstitial lung disease, drug-induced pneumonitis, and autoimmune pneumonitis
* Known active bacterial, viral, fungal, or other infection, or any major episode of infection requiring treatment with IV antibiotics within 4 weeks of Day 1 of Cycle 1
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Known or suspected history of hemophagocytic lymphohistiocytosis
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
* Active Hepatitis B infection
* Active Hepatitis C infection
* Known history of HIV positive status
* History of progressive multifocal leukoencephalopathy (PML)
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Other malignancy that could affect compliance with the protocol or interpretation of results
* Active autoimmune disease requiring treatment
* History of autoimmune disease, including, but not limited to: myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Prior allogeneic stem cell transplantation
* Contraindication to treatment for thromboembolism prophylaxis
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to, significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1 Day 1 or anticipation of a major surgical procedure during the course of the study
* Pregnant or lactating or intending to become pregnant during the study
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) according to 2014 Lugano Response Criteria | From randomization to the first occurrence of disease progression as determined by an independent review committee (IRC) or death from any cause (up to approximately 8.5 years)

SECONDARY OUTCOMES:
PFS as Determined by the Investigator | From randomization to the first occurrence of disease progression or death from any cause (up to approximately 8.5 years)
Complete Response Rate | Up to approximately 8.5 years
Objective Response Rate (ORR) | Up to approximately 8.5 years
Overall Survival (OS) | From randomization to death from any cause (up to approximately 8.5 years)
Duration of Objective Response (DOR) | From the first occurrence of a documented objective response (complete response or partial response) to disease progression or death from any cause, whichever occurs first (up to approximately 8.5 years)
Duration of Complete Reponse (DOCR) | From the first occurrence of a documented CR to disease progression or death from any cause, whichever occurs first (up to approximately 8.5 years)
Time to Deterioration in Physical Functioning and Fatigue, as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) | Up to approximately 8.5 years
Time to Deterioration in Lymphoma Symptoms, as Measured by the Functional Assessment of Cancer Therapy-Lymphoma Subscale (FACT-LymS) | Up to approximately 8.5 years
Percentage of Participants with Adverse Events (AEs) | Up to approximately 8.5 years
Serum Concentration of M + Len | Up to approximately 8.5 years
Area Under the Curve (AUC) of M + Len | Up to approximately 8.5 years
Percentage of Participants with Anti-Drug Antibodies (ADAs) | Up to approximately 8.5 years
Time to New Anti-Lymphoma Treatment (TTNALT) | From randomization to the first documented administration of a new anti-lymphoma treatment (up to approximately 8.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (112):
- United States (17):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Winship Cancer Institute, Atlanta, Georgia
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - Investigative Clinical Research of Indiana, LLC, Noblesville, Indiana
  - Johns Hopkins Uni, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cancer & Hematology Center of West Michigan, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - NYU Long Island Hospital, Mineola, New York
  - NYU Langone Ambulatory Care Center, New York, New York
  - Montefiore Medical Center - Montefiore Medical Park, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Univ Health Svcs, Winston-Salem, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
- Australia (4):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital Woolloongabba, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Geelong Hospital, Geelong, Victoria
- Brazil (4):
  - ICTR Curitiba, Curitiba, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- China (15):
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Cancer Center, Sun Yat-sen University of Medical Sciences, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhejiang Cancer Hospital, Zhejiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- France (18):
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Ch De Chambery, Chambéry
  - Hopital Henri Mondor, Créteil
  - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU Saint Eloi, Montpellier
  - CHU NANTES - Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes - Hôpital Carémeau, Nîmes
  - Hôpital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital De Haut Leveque, Pessac
  - Ch Lyon Sud, Pierre-Bénite
  - Hopital De La Miletrie, Poitiers
  - CHU de Reims, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - ICANS, Strasbourg
- Germany (7):
  - Vivantes Klinikum Am Urban Klinik für Innere Medizin Hämatologie und Onkologie, Berlin
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf, Dresden
  - Universitätsklinikum Halle, Halle
  - Uniklinik Heidelberg, Medizinische Klinik & Poliklinik V, Heidelberg
  - Klinik und Poliklinik f. Innere Medizin III des Universitätsklinikums Regensburg, Regensburg
  - Universitätsklinik Rostock, Rostock
  - Universtitätsklinikum Ulm, Ulm
- Italy (6):
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - U.O. Ematologia AUSL Ravenna, Ravenna, Emilia-Romagna
  - Ospedale V. Cervello, Palermo, Sicily
  - Ospedali Riuniti Umberto I, Ancona, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Ematologia/immunologia Clinica Azienda Ospedaliera Policlinico di Padova, Padua, Veneto
- Japan (8):
  - Aichi Cancer Center, Aichi
  - National Cancer Center Hospital East, Chiba
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Mie University Hospital, Mie
  - Tohoku University Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - Pratia Onkologia Katowice, Katowice
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroc?aw
- Russia (2):
  - City Clinical Botkin's Hospital, Moscow
  - Penza Regional Oncology Dispensary, Penza
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (5):
  - Hospital de Donostia, Guipuzcoa, Guipuzcoa
  - Hospital Universitario la Paz, Madrid
  - Hospital General Universitario J.M Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (4):
  - Chang Gung Medical Foundation - Kaohsiung;Oncology, Kaoisung
  - National Taiwan Universtiy Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Turkey (Türkiye) (4):
  - Hacettepe Uni Medical Faculty, Ankara
  - Atakent Acibadem Private Hosptial Halkali Merkez Mh.,, Istanbul
  - Marmara Ün?Vers?Tes? ?Stanbul Pend?K E??T?M Ve Ara?Tirma Hastanes?, Istanbul
  - Koc Universitesi (KU) Tip Fakultesi (Koc University School of Medicine), Sarıyer
- United Kingdom (5):
  - Royal Cornwall Hospitals NHS Trust, Cornwall
  - Gloucestershire Royal Hospital, Gloucester
  - Hammersmith Hospital, London
  - Nottingham City Hospital, Nottingham
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing